CLINICAL TRIAL: NCT03892694
Title: Characterizing the Mechanism of Action of Metered Cryospray for the Treatment of Patients With Chronic Obstructive Pulmonary Disease With Chronic Bronchitis
Brief Title: Metered Cryospray for the Treatment of Patients With Chronic Obstructive Pulmonary Disease With Chronic Bronchitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 022
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: COPD; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centre, randomised, blinded, sham controlled trial with 1:1 randomisation. Sham-control arm subjects are eligible to receive treatment after the 6-month visit.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Sham controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Active Comparator): MCS
  Interventions: Device: RejuvenAir System
- Sham Control (Sham Comparator): Sham
  Interventions: Other: Sham

INTERVENTIONS:
Device: RejuvenAir System — Bronchial metered cryospray using RejuvenAir® System.
  Arms: Treatment
Other: Sham — Sham control procedure
  Arms: Sham Control

SUMMARY:
To evaluate the relationship between airway structure and function in patients with chronic bronchitis treated with metered cryospray (MCS).

DETAILED DESCRIPTION:
To identify the molecular and cellular targets of MCS treatment and determine the mechanistic relationship to airways remodelling in patients with chronic bronchitis. Phenotype, characterise and correlate clinical, physiological, histological and molecular parameters in patients with chronic bronchitis.

ELIGIBILITY:
Inclusion Criteria:

Each Subject must meet the following criteria to be enrolled in the study:

1. Males and females ≥40 to <80 years of age.
2. Subject is able to read, understand, and sign a written Informed Consent in order to participate in the study.
3. Subject has a diagnosis of CB and COPD and has been symptomatic for a minimum of two years. (Chronic Bronchitis is defined clinically as chronic productive cough for 3 months in each of 2 successive years in a patient in whom other causes of productive cough have been excluded).
4. Subject is classified as having moderate or severe (GOLD stage 2-3) airflow obstruction defined by a post-bronchodilator of =>30% FEV1 to <80% predicted with a baseline FEV1/FVC of <0.70.
5. Subject has a COPD assessment tool (CAT) score of ≥10.
6. Subject is being treated according to current medically accepted treatment guidelines without successful resolution of chronic bronchitis and agrees to continue maintenance pulmonary/COPD medications (as defined per GOLD Standard for medications) for the duration of the study (subject must be on a regime of pulmonary medications for a minimum of 2 weeks prior to enrolment into the study).
7. Smoking history of at least 10 pack years.
8. Non-smoking for a minimum of 2 months prior to consent and agrees to continue not smoking for the duration of the study.
9. Subject is able to adhere to and undergo 4 bronchoscopic procedures (5 for control subjects accepting cross over option), in the opinion of the investigator or per hospital guidelines.
10. For women of childbearing potential: non-pregnant, non-lactating, and agree to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for the duration of the study.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Subject has had an acute pulmonary infection, exacerbation or pneumonia requiring medical treatment (with antibiotics and/or steroids) within 6 weeks of initially planned study bronchoscopy.
2. Diagnosis of asthma with an onset before 30 years of age.
3. Subject has Alpha-1 antitrypsin deficiency.
4. Subject has other origins of respiratory disease aside from chronic bronchitis and COPD.
5. Subject is using e-cigarettes, vaping or taking any oral or inhaled substances not prescribed by a physician.
6. Subject has untreatable or life-threatening arrhythmias, or history of inability to adequately oxygenate during a bronchoscopy, or has acute respiratory failure with hypercapnia.
7. Subject has bullous emphysema characterized as large bullae >30 millimetres on HRCT; or subject has stenosis in the tracheobronchial system, tracheobronchomegaly, trachea-bronchomalacia, amyloidosis or cystic fibrosis.
8. Subject has clinically significant bronchiectasis
9. Subject has had a transplant procedure (any).
10. Subject has a known mucosal tear, has undergone prior lung surgery such as pneumonectomy, lobectomy, bullectomy, or lung volume reduction surgery, bronchial thermoplasty, rheoplasty or cryotherapy.
11. Subject has had a prior lung device procedure, including emphysema stent(s) implanted, lung coils, valves, lung denervation or other devices for emphysema.
12. Subject is unable to temporarily discontinue use of anticoagulant therapy: warfarin, Coumadin, LMWH, heparin, clopidrogel (or equal).
13. Subject has a serious medical condition, such as: uncontrolled coagulopathy or bleeding disorder, congestive heart failure, uncontrolled angina, myocardial infarction in the past year, renal failure, liver disease, cerebrovascular accident within the past 6 months, uncontrolled diabetes, uncontrolled hypertension, autoimmune disease or uncontrolled gastric reflux.
14. Subject has or is receiving chemotherapy or active radiation therapy within the past 6 months or is expected to receive chemotherapy during participation in this study.
15. Subject is or has been in another clinical investigational study within 6 weeks of enrolment.
16. Subject has known sensitivity to medication required to perform bronchoscopy (such as lidocaine, atropine, and benzodiazepines).

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Goblet cell density | 6-months post treatment
  Difference in change relative to baseline in goblet cell density per mm of basement membrane in endobronchial cryobiopsies at 6-months between treatment and sham-control groups

SECONDARY OUTCOMES:
Histopathological examination of endobronchial cryobiopsies to determine Inflammatory cells and subtype density per mm of basement membrane | 6-months post treatment
  Proportion of inflammatory cells per mm of basement membrane for Neutrophil and Lymphocyte sequencing (RNA-seq)
Histopathological examination of endobronchial cryobiopsies to determine epithelial cell density and area (including respiratory epithelial, goblet and basal cells) per mm of basement membrane | 6-months post treatment
  Proportion of epithelial cells per mm of basement membrane for Ciliary and Goblet cells
Transcriptomics: Epithelial gene expression as measured by global gene expression sequencing (RNA-seq) | 6-months post treatment
  Transcriptomics: Epithelial gene expression as measured by global gene expression sequencing (RNA-seq)
Pulmonary function tests including spirometry, body plethysmography and transfer factors KCO and TLCO | 6-months post treatment
  Pulmonary function tests including spirometry, body plethysmography and transfer factors KCO and TLCO
Patient reported outcome measures including SGRQ, mMRC, CAT and Cough Questionnaires | 6-months post treatment
  Patient reported outcome measures including SGRQ, mMRC, CAT and Cough Questionnaires
Health care utilisation assessments including number of respiratory exacerbations, emergency room visits, hospital and intensive care unit admissions related to respiratory adverse events | 6-months post treatment
  Health care utilisation assessments including number of respiratory exacerbations, emergency room visits, hospital and intensive care unit admissions related to respiratory adverse events
The 6-minute walk tests | 6-months post treatment
  The 6-minute walk tests

OTHER OUTCOMES:
Microvesicle quantification | 6-months post treatment
  Microvesicle quantification
Lobar volumes and gas trapping as determined by quantitative CT and parametric response mapping | 6-months post treatment
  Lobar volumes and gas trapping as determined by quantitative CT and parametric response mapping
Small airways function as assessed by Impulse Oscillometry (IOS) | 6-months post treatment
  Small airways function as assessed by Impulse Oscillometry (IOS)
Composition of epithelial ultrastructure as assessed by transmission electron microscopy | 6-months post treatment
  Composition of epithelial ultrastructure as assessed by transmission electron microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Pallav Shah, MD, Principal Investigator — The Royal Brompton Hospital
Locations (2):
- University Medical Center Groningen, Groningen, Netherlands
- The Royal Brompton Hospital, London, United Kingdom